CLINICAL TRIAL: NCT07088250
Title: Statins for Treatment Of Primary IntraCerebral Hemorrhage (STOP ICH)
Brief Title: Statins for Treatment of Primary Intracerebral Hemorrhage
Acronym: STOP ICH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Qi Li, Professor, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YX2023-041(F1)
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Cerebrovascular Disorders; Intracranial Hemorrhages; Intracranial Hemorrhage; Intracerebral Haemorrhage
Keywords: Intracerebral hemorrhage; Treatment; Atorvastatin; Outcome
MeSH Terms: conditions — Cerebrovascular Disorders; Intracranial Hemorrhages; Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin Treatment plus Best Medical Treatment (Experimental): Patients in this group will receive atorvastatin treatment plus best medical treatment.
  Interventions: Drug: Atorvastatin Treatment; Other: Best Medical Treatment
- Best Medical Treatment (Active Comparator): Patients in this group will receive best medical treatments in accordance with the guideline-directed management for ICH.
  Interventions: Other: Best Medical Treatment

INTERVENTIONS:
Drug: Atorvastatin Treatment — Atorvastatin 20 mg once daily for 21 days.
  Arms: Atorvastatin Treatment plus Best Medical Treatment
Other: Best Medical Treatment — Patients in this group will receive best medical treatments in accordance with the guideline-directed management for ICH.

SUMMARY:
The STOP ICH trial is a multicenter, prospective, randomized, open-label, blinded end-point (PROBE) study designed to assess the efficacy and safety of atorvastatin in patients with intracerebral hemorrhage (ICH) presenting within 3 to 24 hours of symptom onset.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, randomized, open-label, blinded end-point (PROBE) clinical trial aimed at evaluating the efficacy and safety of atorvastatin in patients with spontaneous intracerebral hemorrhage (ICH). Eligible participants include adults aged 18 to 80 years presenting with spontaneous ICH who are enrolled within 3 to 24 hours from symptom onset or the last known well time, provided they meet all inclusion criteria and no exclusion criteria. A total of 264 patients will be randomized in a 1:1 ratio into two treatment arms: the control group, receiving best medical treatment (BMT) in accordance with current ICH guidelines, and the experimental group, receiving BMT plus atorvastatin at a dosage of 20 mg once daily for 21 consecutive days. The primary objective is to determine whether atorvastatin improves clinical outcomes in patients with ICH. The primary efficacy endpoint is the proportion of patients with a poor functional outcome at 90 days, defined as a modified Rankin Scale (mRS) score of 4 to 6.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of spontaneous intracerebral hemorrhage (ICH) confirmed by computed tomography (CT);
* Age 18-80 years;
* Hematoma located in the supratentorial region;
* Time from symptom onset or last known well to baseline CT ranging from 3 to 24 hours;
* Atorvastatin treatment can be initiated within 48 hours of symptom onset or last known well;
* Glasgow Coma Scale (GCS) score ≥9;
* Baseline hematoma volume of 5-35 mL;
* Signed informed consent obtained.

Exclusion Criteria:

* ICH secondary to trauma, tumor, aneurysm, arteriovenous malformation (AVM), vascular anomaly, hemorrhagic transformation of infarction, cerebral venous thrombosis, or anticoagulant-related ICH;
* Patients who have undergone or are scheduled for immediate surgical intervention;
* Pregnancy or lactation;
* Use of oral anticoagulants within 1 month prior to symptom onset;
* Pre-stroke mRS >1;
* Known allergy to statins, active liver disease, liver dysfunction, or rhabdomyolysis;
* Known terminal illness with a pre-stroke life expectancy of less than three months, or patients with planned withdrawal of care.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-05-06 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Poor functional outcome | 90 ± 7 days
  The proportion of poor functional outcome, defined as a modified Rankin Scale (mRS) score of 4-6 at 90 ± 7 days. The mRS is a widely used 6-point scale for assessing disability and functional outcomes after stroke, where higher scores represent worse outcomes.

SECONDARY OUTCOMES:
Functional independence | 90 ± 7 days
  The proportion of functional independence, defined as a modified Rankin Scale (mRS) score of 0-2 at 90 ± 7 days. The mRS is a widely used 6-point scale for assessing disability and functional outcomes after stroke, where higher scores represent worse outcomes.
Ordinal distribution of mRS | 90 ± 7 days
  Ordinal distribution of the modified Rankin Scale (mRS) at 90 ± 7 days. The mRS is a widely used 6-point scale for assessing disability and functional outcomes after stroke, where higher scores represent worse outcomes
Changes in hematoma volume from baseline to 24 ± 12 hours | 24 ± 12 hours
  Absolute and relative changes in hematoma volume, measured as the difference between baseline CT scan and follow-up CT scan performed at 24 ± 12 hours post-baseline.
Changes in hematoma volume from baseline to 7 ± 1 days | 7 ± 1 days
  Absolute and relative changes in hematoma volume, measured as the difference between baseline CT scan and follow-up CT scan performed at 7 ± 1 days post-baseline.
Changes in hematoma volume from 24 ± 12 hours to 7 ± 1 days | between 24 ± 12 hours and 7 ± 1 days
  Absolute and relative changes in hematoma volume, measured as the difference between 24 ± 12 hours CT scan and 7 ± 1 days CT scan.
Changes in perihematomal edema (PHE) volume from baseline to 7 ± 1 days | 7 ± 1 days
  Changes in PHE volume, measured as the difference between baseline CT scan and follow-up CT scan performed at 7 ± 1 days post-baseline.
Changes in perihematomal edema (PHE) volume from 24 ± 12 hours to 7 ± 1 days | 7 ± 1 days
  Changes in PHE volume, measured as the difference between 24 ± 12 hours CT scan and 7 ± 1 days CT scan

OTHER OUTCOMES:
Recurrent intracerebral hemorrhage | 90 ± 7 days
  The incidence of recurrent intracerebral hemorrhage within 90 ± 7 days
All cause mortality | 90 ± 7 days
  All cause mortality at 90 ± 7 days.
Any adverse event/serious adverse event | 90 ± 7 days
  Any adverse events or serious adverse events occurred within 90 ± 7 days

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Anqing First People's Hospital of Anhui Province, Anqing, Anhui
  - Fuyang City Sixth People's Hospital, Fuyang, Anhui
  - Fuyang Hospital of Anhui Medical University, Fuyang, Anhui
  - Fuyang People's Hospital, Fuyang, Anhui
  - Hefei Eighth People's Hospital, Hefei, Anhui
  - Hefei First People's Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Huainan Xinhua Hospital, Huainan, Anhui
  - The First Affiliated Hospital of Anhui University of Science and Technology (Huainan First People's Hospital), Huainan, Anhui
  - Huoqiu First People's Hospital, Lu'an, Anhui
  - Shucheng People's Hospital, Lu'an, Anhui
  - Si County People's Hospital, Suzhou, Anhui
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Kaifeng Central Hospital, Kaifeng, Henan
  - Xihua County People's Hospital, Zhoukou, Henan
  - Xiangyang Hospital of Traditional Chinese Medicine, Xiangyang, Hubei
  - The First People's Hospital of Chenzhou, Chenzhou, Hunan
  - Yancheng First People's Hospital, Yancheng, Jiangsu
  - Chengdu Western Hospital, Chengdu, Sichuan
  - Panzhihua Central Hospital, Panzhihua, Sichuan
  - Dazhu County People's Hospital, Dazhou, Sizhuan
  - The Third Affiliated Hospital of Chong Qing Medical University, Chongqing

IPD SHARING:
Plan to Share IPD: Undecided